CLINICAL TRIAL: NCT00498394
Title: Effects of a Ketogenic Diet on Body Weight and Cardiovascular Risk Factors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: American Heart Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0060334B
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Diet fads
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Clinical diet trial

SUMMARY:
This pilot study is a randomized, controlled clinical trial to compare anthropometric and metabolic changes associated with six months of weight management by means of a very low carbohydrate diet or a calorically-restricted low fat diet. We hypothesized that the low fat diet would be associated with more weight loss and improvement of cardiovascular risk factors than the low carbohydrate diet.

DETAILED DESCRIPTION:
Low carbohydrate diets, including high-fat, 'ketogenic' diets, have moved to the forefront of popular diets promoted for weight loss in the United States. These diet plans have been aggressively marketed to millions of Americans every year. However, there has been virtually no rigorous study of low carbohydrate, high fat diets either with regard to efficacy in promoting weight loss or effects on cardiovascular risk factors. Because very low carbohydrate diets (i.e., the ketogenic diets) recommend increased intake of fat, and saturated fat, we hypothesized that following one of these diet plans could actually worsen important risk factors for cardiovascular disease. This is an issue of great importance because large numbers of people experiment with low carbohydrate diets despite not knowing their effects on blood pressure, plasma lipid levels, and glucose tolerance. Therefore, we have proposed a clinical trial to test our hypothesis. In this study, we will compare the effects of three months of a ketogenic diet (as promoted by Dr. Robert Atkins) with three months of a weight loss diet that conforms to the American Heart Association dietary guidelines in a group of 100 otherwise healthy obese subjects. During the course of the study, we will determine the effects of diet on 1) body weight, percent fat, and resting metabolic rate, 2) blood pressure, 3) plasma lipids, 4) measures of glucose tolerance, and 5) measures of psychological health and eating behaviors. This pilot study will provide the preliminary data needed to demonstrate the efficacy (or lack thereof) of a popular weight loss technique (i.e., the ketogenic diet) that is currently being criticized by professional organizations. Armed with preliminary data, the investigators plan to further investigate the long-term anthropometric and metabolic effects of ketogenic diets with a larger sample.

ELIGIBILITY:
Inclusion Criteria:

* Obese men and women with a BMI of 30-34 kg/m2, at least 18 years of age, who have had stable body weight (i.e., no gain or loss of >5% of body weight) for the preceding six months, who have normal oral glucose tolerance, and who are able to commit to a six month study.

Exclusion Criteria:

* Pregnancy, lactation, active medical or mental illness requiring treatment, recent (within 1 year) use of appetite suppressing compounds, previous use of the ketogenic diet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2000-06; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 months

SECONDARY OUTCOMES:
Body fat via dual energy x-ray absorptiometry (DXA) | 6 months
Resting metabolic rate via indirect calorimetry | 6 months
Blood pressure | 6 months
Fasting plasma total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides | 6 months
Fasting insulin and glucose | 6 months
Psychological health and eating behaviors via surveys | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J Brehm, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Brehm BJ, Seeley RJ, Daniels SR, D'Alessio DA. A randomized trial comparing a very low carbohydrate diet and a calorie-restricted low fat diet on body weight and cardiovascular risk factors in healthy women. J Clin Endocrinol Metab. 2003 Apr;88(4):1617-23. doi: 10.1210/jc.2002-021480. PMID 12679447
- [Result] Brehm BJ, Spang SE, Lattin BL, Seeley RJ, Daniels SR, D'Alessio DA. The role of energy expenditure in the differential weight loss in obese women on low-fat and low-carbohydrate diets. J Clin Endocrinol Metab. 2005 Mar;90(3):1475-82. doi: 10.1210/jc.2004-1540. Epub 2004 Dec 14. PMID 15598683
- [Result] O'Brien KD, Brehm BJ, Seeley RJ, Bean J, Wener MH, Daniels S, D'Alessio DA. Diet-induced weight loss is associated with decreases in plasma serum amyloid a and C-reactive protein independent of dietary macronutrient composition in obese subjects. J Clin Endocrinol Metab. 2005 Apr;90(4):2244-9. doi: 10.1210/jc.2004-1011. Epub 2005 Jan 25. PMID 15671108